CLINICAL TRIAL: NCT05364424
Title: A Phase IB, Open-Label, Multicenter, Single Arm Study Evaluating the Preliminary Efficacy, Safety, and Pharmacokinetics of Glofitamab in Combination With Rituximab Plus Ifosfamide, Carboplatin Etoposide Phosphate in Patients With Relapsed/Refractory Transplant or CAR-T Therapy Eligible Diffuse B-Cell Lymphoma
Brief Title: A Study Evaluating the Efficacy, Safety, and Pharmacokinetics of Glofitamab in Combination With Rituximab Plus Ifosfamide, Carboplatin Etoposide Phosphate in Participants With Relapsed/Refractory Transplant or CAR-T Therapy Eligible Diffuse B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO43693
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab; obinutuzumab; tocilizumab; Rituximab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- R/R DLBCL (Experimental): Participants will receive up to 3 21-day cycles of glofitamab, rituximab, ifosfamide, carboplatin, and etoposide (glofit-R-ICE).
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Tocilizumab; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Glofitamab — Participants will receive intravenous (IV) glofitamab for up to 3 cycles.
Drug: Obinutuzumab — Participants will receive IV obinutuzumab on Cycle 1 Day 1.
Drug: Tocilizumab — Participants will receive IV tocilizumab as necessary to manage cytokine release syndrome (CRS) events.
Drug: Rituximab — Participants will receive up to 2 doses of IV rituximab.
Drug: Ifosfamide — Participants will receive IV ifosfamide for up to 3 cycles.
Drug: Carboplatin — Participants will receive IV carboplatin for up to 3 cycles.
Drug: Etoposide — Participants will receive IV etoposide for up to 3 cycles.

SUMMARY:
The purpose of this study is to evaluate the preliminary efficacy, safety, and pharmacokinetics of glofitamab (glofit) in combination with rituximab plus ifosfamide, carboplatin, and etoposide (R-ICE) in participants with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL), who have failed one prior line of therapy incorporating an anti-cluster of differentiation (CD) 20 antibody (i.e., rituximab) and an anthracycline, and who are transplant or chimeric antigen receptor T-cell (CAR-T) therapy eligible, defined as being medically eligible for intensive platinum-based salvage therapy followed by autologous stem cell transplantation (ASCT) or for CAR-T therapy.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy ≥ 12 weeks
* Histologically confirmed B-cell lymphoma
* One line of prior systemic therapy including an anti-CD20 monoclonal antibody (i.e. rituximab) and an anthracycline
* Relapsed or refractory disease after first-line chemoimmunotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Participant must be a candidate for high-dose chemotherapy followed by ASCT or CAR-T therapy

Exclusion Criteria:

* Treatment with more than one prior line of therapy for DLBCL
* Primary mediastinal B-cell lymphoma
* Prior treatment with glofitamab or other bispecific antibodies targeting both CD20 and CD3
* Peripheral neuropathy assessed to be Grade > 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 at enrollment
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to first study treatment
* Treatment with monoclonal antibodies for the purposes of treating cancer within 4 weeks prior to first study treatment
* Primary or secondary CNS lymphoma at the time of enrollment or history of CNS lymphoma
* Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Known history of progressive multifocal leukoencephalopathy
* Adverse events from prior anti-cancer therapy that have not resolved to Grade 1 or better (with the exception of alopecia and anorexia, or as otherwise permitted by inclusion criteria)
* Prior solid organ transplantation
* Prior allogeneic stem cell transplant
* Prior ASCT for lymphoma
* Prior autologous stem cell transplant for any indication other than lymphoma, within 5 years from the start of study treatment
* Active autoimmune disease requiring treatment
* Prior treatment with systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents), within 4 weeks prior to first dose of study treatment
* Ongoing corticosteroid use > 30 mg/day of prednisone or equivalent. Participants who received corticosteroid treatment with ≤ 30 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to Cycle 1 Day 1. Participants may have received a brief (≤ 7 days) course of systemic steroids (≤ 100 mg prednisone equivalent per day) prior to initiation of study therapy for control of lymphoma-related symptoms
* Recent major surgery (within 4 weeks before the first study treatment) other than for diagnosis
* Clinically significant history of cirrhotic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR), defined as the proportion of participants that achieves a CR or PR within three cycles of glofit-R-ICE, as determined by the investigator according to Lugano criteria | Up to 2.5 years

SECONDARY OUTCOMES:
Event-free survival (EFS) after enrollment | From enrollment to the first occurrence of disease progression, initiation of new anti-lymphoma therapy (not including planned ASCT or CAR-T therapy), or death from any cause (whichever occurs first) (up to 2.5 years)
Progression-free survival (PFS) after enrollment | From enrollment to the first occurrence of disease progression or death from any cause (whichever occurs first) as determined by the investigator according to Lugano criteria (up to 2.5 years)
Mobilization-adjusted response rate (MARR) | Up to 2.5 years
  The proportion of participants treated with intent to proceed to ASCT that achieves a CR or PR within three cycles of glofit-R-ICE, as determined by the investigator according to Lugano criteria, and additionally achieves mobilization of a minimum of 2,000,000 CD34+ hematopoietic stem cells/kg for ASCT
Overall survival (OS) after enrollment | From enrollment to death from any cause (up to 2.5 years)
CR rate after enrollment, defined as the proportion of participants that achieves a CR within three cycles of glofit-R-ICE, as determined by the investigator according to Lugano criteria | Up to 2.5 years
Duration of Response (DOR) | From the first occurrence of a documented objective response (CR or PR) to disease progression or death from any cause (whichever occurs first) as determined by the investigator according to Lugano criteria (up to 2.5 years)
Duration of complete response (DOCR) | From the first occurrence of a documented complete response to disease progression or death from any cause (whichever occurs first) as determined by the investigator according to Lugano criteria (up to 2.5 years)
Percentage of participants with adverse events (AEs) | Up to 2.5 years
Percentage of participants with cytokine release syndrome (CRS) | Up to 2.5 years
Maximum serum concentration (Cmax) of glofitamab | Up to 2.5 years
Minimum serum concentration (Cmin) of glofitamab | Up to 2.5 years
Percentage of participants with anti-drug antibodies (ADAs) | From baseline up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (9):
  - Chao Family Comprehensive Cancer Center UCI, Orange, California
  - Memorial Cancer Institute at Memorial West, Pembroke Pines, Florida
  - The University of Chicago, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - New York University Langone Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No